CLINICAL TRIAL: NCT06432504
Title: Variation in the Impact of Coffee on the Metabolic Rate
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shenzhen Institutes of Advanced Technology ,Chinese Academy of Sciences (Other)
Responsible Party: Principal Investigator, John R. Speakman, Professor, Shenzhen Institutes of Advanced Technology ,Chinese Academy of Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: SIAT IRB 221115H0629
Record Dates: First submitted 2024-04-02; First posted 2024-05-29 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Healthy
Keywords: Coffee; Caffeine; Metabolic rate; Caffeine clearance

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- caffeine content 100mg (Experimental): The participants will drink 180 mls coffee
  Interventions: Other: Caffeine content
- caffeine content 200mg (Experimental): The participants will drink 180 mls coffee.
  Interventions: Other: Caffeine content
- caffeine content 300mg (Experimental): The participants will drink 180 mls coffee
  Interventions: Other: Caffeine content
- 13C3 caffeine content 100mg (Experimental): The participants will drink 180 mls coffee (caffeine content 100mg) containing 13C labelled caffeine to trace the pattern of caffeine degradation.
  Interventions: Other: Caffeine content

INTERVENTIONS:
Other: Caffeine content — Participants will drink the same volume of coffee with different amounts of caffeine.

SUMMARY:
The purpose of this study is to explore variation in the impact of coffee on metabolic rate. The investigators plan to recruit healthy participants, half male and half female.

DETAILED DESCRIPTION:
The investigators will study the variation in the impact of coffee on metabolic rate and investigate the impacts of age, sex, body composition and regularity of habitual coffee consumption on this effect. The investigators will recruit healthy participants, half male and half female. Participants will be required to perform no strenuous exercise for 14 hours and no moderate of vigorous exercise for 2 hours before the measurements. When the participants arrive at the lab on the day of the experiment, they will sign an informed consent form, a health history questionnaire and a daily coffee consumption questionnaire. Participants will be randomly allocated into 3 groups and given 180mls of coffee to consume containing 100, 200 or 300 mg of caffeine. A fourth group will be dosed with 100 mg of caffeine containing 13C uniform labelled caffeine to trace the pattern of caffeine degradation via the appearance of 13CO2 in the breath and labelled compounds in the urine. The primary outcome is the change in resting metabolic rate from before and after coffee drinking. Secondary outcome measures are heart rate, electrocardiogram, blood pressure, body temperature which will be measured before and after the coffee consumption. Professional nurses will take 8ml of venous blood from all participants as genotyping blood samples. Genomic DNA will be extracted from whole blood samples and analysed for single nucleotide polymorphisms (SNPS).

ELIGIBILITY:
Inclusion Criteria:

Healthy adults 18-40 years old

Exclusion Criteria:

Those who have undergone surgery in the past 6 months. People are requiring long-term medication. People have metabolic diseases, like diabetes, hypoglycemia, gout, osteoporosis, etc.

People have digestive diseases, like gastric ulcer, pancreatitis, intestinal obstruction, etc.

Those who have recently lost weight for various medical reasons ( like cancer, etc.).

People are suffering from infectious diseases ( like HIV, etc.). People have blood phobia, pathological hypo or hyper tension. People with impaired glucose tolerance. Those who are afflicted with claustrophobia.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-03-06 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Resting energy expenditure | On the first moring of experiment, it lasts 0.5 hours and 3 hours.
  Resting energy expenditure will be measured using indirect calorimetry via a respiratory hood system (COSMED). The subject attends in the lab after an overnight fast. The person lies down on a flat bed and the hood is placed over their head. Resting energy expenditure will be measured before and after coffee consumption.
  The extra energy expenditure is equal to the resting energy expenditure after drinking coffee minus the resting energy expenditure before drinking coffee.
Urine metabolites | On the first moring of experiment, it lasts 0.5 hours and 3 hours.
  The contents of metabolites will be measured by gas chromatography-mass spectrometry (GC-MS) and liquid chromatography-mass spectrometry (LC-MS ).
Expired gases | On the first moring of experiment, it lasts 0.5 hours and 3 hours.
  Gases will be collected before and after coffee consumption, Gases will be measured by CO2 isotope analyzer (CCIA2-912) to observe the change of labelled CO2.

SECONDARY OUTCOMES:
Body temperature | On the first moring of experiment, it lasts 0.5 hours and 3 hours.
  Body temperature of participants will be measured by body temperature patch (RIT-P02-MED) before and after coffee consumption.
Electrocardiogram (ECG) | On the first moring of experiment, it lasts 0.5 hours and 3 hours.
  ECG of participants will be measured by Amu ECG belt before and after coffee consumption, the changes in P wave, PR interval, PR segment, QRS wave group, J point, ST segment, T wave, QT interval, and U wave will be observe.
Blood samples | Baseline : empty stomach On the first moring of experiment.
  Venous blood collected by nurses, blood samples will be used for whole genome exon sequencing to analyze single nucleotide polymorphisms.
Blood pressure | On the first moring of experiment, it lasts 0.5 hours and 3 hours.
  Systolic and diastolic blood pressure of participants will be measured by Omron digital sphygmomanometer before and after coffee consumption.
Height | On the first moring of experiment, it lasts 5 minutes.
  Height will be measured by seca 217 stable stadiometer.
Body weight | On the first moring of experiment, it lasts 5 minutes.
  Fasting body weight will be measured by Bioimpedance Analysis (TANITA, MC-980).
Fat mass | On the second moring of experiment, it lasts 10 minutes.
  Fat mass will be measured by Magnetic Resonance Imaging (Shanghai united imaging, uMR 790 ).
Fat free mass | On the first moring of experiment, it lasts 5 minutes.
  Fat free mass will be Bioimpedance Analysis (TANITA, MC-980).
Bone mass | On the first moring of experiment, it lasts 10 minutes.
  Bone mass will be measured by Dual Energy X-ray Absorptiometry (Horizon Wi).
Heart rate | On the first moring of experiment, it lasts 0.5 hours and 3 hours.
  Heart rate will be measured by Omron sphygmomanometer.
Body water, extracellular fluid and intracelluar fluid | On the first moring of experiment, it lasts 0.5 hours and 3 hours.
  Body water, extracellular fluid and intracelluar fluid will be measured by Bioimpedance Analysis (TANITA, MC-980).

CONTACTS AND LOCATIONS:
Overall Officials: John R Speakman, PhD, Study Chair — Shenzhen Institutes of Advanced Technology ,Chinese Academy of Sciences
Locations (1):
- Shenzhen Institute of Advanced Technology, Shenzhen, Guangdong, China